CLINICAL TRIAL: NCT05943769
Title: The Impact of Root End Filling Material Type and the Application of Bone Graft on Healing of Periapical Tissues After Endodontic Microsurgery (A Clinical Randomized Controlled Trial)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FDASU-RecID041910
Record Dates: First submitted 2023-07-06; First posted 2023-07-13 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-06

CONDITIONS: Periapical Diseases; Periapical Cyst
Keywords: Apicoectomy; Bone graft; Endodontic surgery; MTA; TotalFill; Apical lesions
MeSH Terms: conditions — Periapical Diseases; Radicular Cyst | interventions — Apicoectomy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- MTA (Experimental): Root end filling material is MTA without bone graft in the defect.
  Interventions: Procedure: Apical microsurgery
- TotalFill (Experimental): Root end filling material is TotalFill without bone graft in the defect.
  Interventions: Procedure: Apical microsurgery
- MTA & bone (Experimental): Root end filling material is MTA with the addition of composite bone graft in the defect.
  Interventions: Procedure: Apical microsurgery
- TotalFill & bone (Experimental): Root end filling material is TotalFill with the addition of composite bone graft in the defect.
  Interventions: Procedure: Apical microsurgery

INTERVENTIONS:
Procedure: Apical microsurgery — inoculation of the periapical or the periradicular lesion with the sectioning of the apical 3mm of the root followed by root-end cavity preparation and retro-filling with the MTA or TotalFill with or without composite bone grafting according to patient allocation.
  Other Names: apicoectomy

SUMMARY:
The goal of this triple blinded randomized clinical trial is to evaluate the effect of combining different bioactive root end filling materials with composite bone graft (xenogeneic mixed with autogenous bone fragments) on the healing process of periapical tissues after endodontic micro-surgery procedure on patients with small to moderate sized lesions. The main questions it aims to answer are:

Will the use of Totalfill in Endodontic surgeries show comparable results to the gold standard MTA? Will the addition of composite bone graft (Xenogenic and Autogenous) affect the healing of small to moderate sized lesions? Is there any interaction between composite bone graft and different bioactive root-end filling materials? Participants were allocated to 4 different groups according to the root-end filling material used with or without bone graft.

Reseachers compared between MTA only group, Totalfill only group, MTA with bone group, and Totalfill with bone group to evaluate healing of the periapical lesion using CBCT after 12 months follow up period.

ELIGIBILITY:
Inclusion Criteria:

All patients must be medically free from any systemic disease that can affect bone healing.

Age range of the patient should be between 20 - 45 years old. All patients must have good oral hygiene. The size of the radiolucent area is of small-moderate size (up to 3 cm in highest diameter at any axis in CBCT), related to a single rooted maxillary tooth.

Periradicular disease in a root-filled tooth where orthograde root canal treatment options has failed,

Exclusion Criteria:

Patient with systemic disease that may affect bone healing. Patients above 45 years or patients below 20 years. Patients with very poor oral hygiene. Teeth presenting with apico-marginal defects or teeth with periodontal disease (periodontal pockets and/or mobility).

Surgery after previous endodontic surgery (re-surgery cases), root resections and amputations, cases presenting with root fractures.

Patients with history of allergies to any of the medications to be used during or after the surgery.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Healing | 12 months
  Assessing healing using CBCT

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams univetsity, Cairo, Egypt